CLINICAL TRIAL: NCT04962022
Title: COVID-19: A PHASE 1, OPEN-LABEL, FIXED SEQUENCE, 2-PERIOD CROSSOVER STUDY TO ESTIMATE THE EFFECT OF ITRACONAZOLE ON THE PHARMACOKINETICS OF PF-07321332/RITONAVIR IN HEALTHY PARTICIPANTS
Brief Title: Drug-Drug Interaction Study Assessing Effect of Itraconazole on PF-07321332/Ritonavir in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: C4671015; 2021-003308-42 (EudraCT Number)
Record Dates: First submitted 2021-07-10; First posted 2021-07-14 (Actual); Results first posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2022-08

CONDITIONS: Healthy Participant
Keywords: Drug-drug interaction; Itraconazole; CYP3A4 inhibitor
MeSH Terms: interventions — nirmatrelvir and ritonavir drug combination; Itraconazole

STUDY DESIGN:
Intervention Model Description: This is a Phase I, fixed sequence, 2-period study to evaluate the effect of the strong CYP3A4 inhibitor, itraconazole, on the PK of PF-07321332 and ritonavir in healthy participants. A total of 12 healthy participants will be enrolled into this study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Period 1 (Experimental): PF-07321332/ritonavir orally
  Interventions: Drug: PF-07321332/ritonavir
- Period 2 (Experimental): Itraconazole + PF-07321332/ritonavir orally.
  Interventions: Drug: Itraconazole; Drug: PF-07321332/ritonavir

INTERVENTIONS:
Drug: PF-07321332/ritonavir — Administered orally every 12 hours for days for a total of 5 doses from Day 1 through Day 3
  Arms: Period 1
Drug: Itraconazole — Administered orally once daily for 8 days from Days 1 through 8
  Arms: Period 2
Drug: PF-07321332/ritonavir — Administered orally BID for 3 day for a total on 5 doses starting on Day 4 through Day 6
  Arms: Period 2

SUMMARY:
The purpose of this study is to estimate the effect of a strong inhibitor of CYP3A4 (itraconazole) on the pharmacokinetics (PK) of PF-07321332/ritonavir in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants who are overtly healthy as determined by medical evaluation including medical history, PE, laboratory tests, vital signs and standard 12 lead ECGs.
2. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
3. Female participants must have a negative pregnancy test.
4. BMI of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb). -

Exclusion Criteria:

1. Positive test result for SARS-CoV-2 infection at the time of Screening or Day -1.
2. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
3. Clinically relevant abnormalities requiring treatment (eg, acute myocardial infarction, unstable ischemic conditions, evidence of ventricular dysfunction, serious tachy or brady arrhythmias) or indicating serious underlying heart disease (eg, prolonged PR interval, cardiomyopathy, heart failure greater than NYHA 1, underlying structural heart disease, Wolff Parkinson-White syndrome).
4. Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
5. History of HIV infection, hepatitis B, or hepatitis C; positive testing for HIV, HBsAg, or HCVAb. Hepatitis B vaccination is allowed.
6. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions or situations related to COVID-19 pandemic (eg, contact with positive case, residence, or travel to an area with high incidence) that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Brussels Clinical Research Unit, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4671015

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a 2-period,fixed-sequence crossover study. A total of 12 participants were assigned to and received the treatment in period 1. One participant discontinued due to withdrawal. The remaining 11 participants completed Period 1 and continued to receive the treatment in Period 2 and all completed Period 2.
Groups:
- PF-07321332 (Suspension)/Ritonavir 300/100 mg BID, Fasted: Participants received PF-07321332/ritonavir 300/100 mg administered orally every 12 hours for a total of 5 doses, from Day 1 morning to Day 3 morning of Period 1.
- Itraconazole 200 mg QD + PF-07321332(Suspension)/Ritonavir 300/100 mg BID, Fasted: Participants received itraconazole 200 mg orally once a day from Days 1 through 8 of Period 2, for a total of 8 doses; and PF-07321332/ritonavir 300/100 mg administered orally every 12 hours from Days 4 through 6 of Period 2, for a total of 5 doses.
Period: Period 1
Arm/Group | PF-07321332 (Suspension)/Ritonavir 300/100 mg BID, Fasted | Itraconazole 200 mg QD + PF-07321332(Suspension)/Ritonavir 300/100 mg BID, Fasted
Started | 12 | 0
Completed | 11 | 0
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Period 2
Arm/Group | PF-07321332 (Suspension)/Ritonavir 300/100 mg BID, Fasted | Itraconazole 200 mg QD + PF-07321332(Suspension)/Ritonavir 300/100 mg BID, Fasted
Started | 0 | 11
Completed | 0 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all participants enrolled in the study.
Groups:
- Overall Study: All participants who received PF-07321332 (suspension)/ritonavir 300/100 mg, Itraconazole 200 mg and PF-07321332(suspension)/ritonavir 300/100 mg in Period 1 and 2, respectively.
Arm/Group | Overall Study
Number analyzed (Participants) | 12
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 0
  18-25 years | 0
  26-35 years | 5
  36-45 years | 3
  >45 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Concentration (Cmax) of PF-07321332
Description: The Cmax of PF-07321332 in the study was observed directly from data.
Time Frame: Days 1, 2, 3 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, and 48 hours postdose on Day 3) in Period 1; Days 1, 4, 5, 6 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48, and 72 hours postdose on Day 6) of Period 2.
Population: The analysis population included all participants who took at least 1 dose of study intervention and in whom at least 1 concentration value was reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-07321332 (Suspension)/Ritonavir 300/100 mg BID, Fasted | Itraconazole 200 mg QD + PF-07321332(Suspension)/Ritonavir 300/100 mg BID, Fasted
Number analyzed (Participants) | 11 | 11
ng/mL | 4678 (17) | 5546 (15)
Statistical Analysis 1: Comparison: PF-07321332 (Suspension)/Ritonavir 300/100 mg BID, Fasted vs Itraconazole 200 mg QD + PF-07321332(Suspension)/Ritonavir 300/100 mg BID, Fasted; Test type: Other — PF-07321332/ritonavir administered alone was the Reference treatment and PF-07321332/ritonavir co-administered with itraconazole was the Test treatment; p = 0.05, Mixed Models Analysis; Specified in comments = 118.57, 90% CI 2-sided [112.50 to 124.97] — Mixed Model was fitted to obtain: 1.Ratio of geometric means 2.90% CI of ratio of geometric means

2. Primary Outcome: Area Under the Plasma Concentration-time Profile From Time Zero to Time Tau (τ), Where Tau=12-hour Dosing Interval(AUCtau) for PF-07321332
Description: The AUCtau of PF-07321332 was determined by Linear/Log trapezoidal method.
Time Frame: as for outcome 1
Population: The analysis population included all participants who took at least 1 dose of study intervention and in whom at least 1 of the PK parameters of interest were reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-07321332 (Suspension)/Ritonavir 300/100 mg BID, Fasted | Itraconazole 200 mg QD + PF-07321332(Suspension)/Ritonavir 300/100 mg BID, Fasted
Number analyzed (Participants) | 11 | 11
ng*hr/mL | 33350 (20) | 46290 (18)
Statistical Analysis 1: Comparison: PF-07321332 (Suspension)/Ritonavir 300/100 mg BID, Fasted vs Itraconazole 200 mg QD + PF-07321332(Suspension)/Ritonavir 300/100 mg BID, Fasted; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.05, Mixed Models Analysis; Specified in comments = 138.82, 90% CI 2-sided [129.25 to 149.11] — Mixed Model was fitted to obtain: 1.Ratio of geometric means 2.90% CI of ratio of geometric means

3. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An Adverse event (AE) was any untoward medical occurrence in a participant. A serious AE was any untoward medical occurrence at any dose that resulted in death; was life-threatening; required hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth, was a suspected transmission via a Pfizer product of an infectious agent,pathogenic or non-pathogenic, was considered serious. The focus of AE summaries was on treatment-emergent AE (TEAE). An AE was considered TEAE if the event occurred during the on-treatment period.
Time Frame: Screening up to Day 35
Population: The analysis population included all participants who took at least 1 dose of study intervention. Participants was analyzed according to the product they actually received.
Measure: Count of Participants; unit: Participants
Groups:
- PF-07321332 (Suspension)/Ritonavir 300/100 mg BID, Fasted: Participants received PF-07321332/ritonavir 300/100 mg administered orally every 12 hours for a total of 5 doses, from Day 1 morning to Day 3 morning in Period 1.
- Itraconazole 200 mg QD + PF-07321332(Suspension)/Ritonavir 300/100 mg BID, Fasted: Participants received itraconazole 200 mg orally once a day from Days 1 through 8 of Period 2; and PF-07321332/ritonavir 300/100 mg administered orally every 12 hours from Days 4 through 6 of Period 2, for a total of 5 doses.
Arm/Group | PF-07321332 (Suspension)/Ritonavir 300/100 mg BID, Fasted | Itraconazole 200 mg QD + PF-07321332(Suspension)/Ritonavir 300/100 mg BID, Fasted
Number analyzed (Participants) | 12 | 11
Participants
  Participants with TEAEs | 7 | 10
  Participants with serious TEAEs | 0 | 0

4. Secondary Outcome: Number of Participants With Laboratory Abnormalities (Without Regard to Baseline Abnormality)
Description: Safety laboratory assessments included urinalysis, hematology, chemistry and other. All the safety laboratory samples were collected following at least a 4-hour fast.
Time Frame: Screening up to Day 9 of Period 2 or Early termination/discontinuation.
Population: The analysis population included all participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07321332 (Suspension)/Ritonavir 300/100 mg BID, Fasted | Itraconazole 200 mg QD + PF-07321332(Suspension)/Ritonavir 300/100 mg BID, Fasted
Number analyzed (Participants) | 12 | 11
Participants
  Monocytes/Leukocytes（%）> 1.2 ✖ ULN | 1 | 2
  Bicarbonate(mEq/L) > 1.1 ✖ ULN | 6 | 0
  Fibrinogen(mg/dl) > 1.25 ✖ Baseline | 0 | 1
  Leukocyte Esterase >= 1 | 0 | 1

5. Secondary Outcome: Number of Participants With Clinically Significant 12-lead Electrocardiogram (ECG) Findings
Description: Triplicate 12-lead ECG readings approximately 2 minutes apart were taken at each test. All ECG assessments were made after at least a 5-minute rest in a supine position and prior to any blood draws or vital sign measurements.
Time Frame: Screening up to Day 9 of Period 2 or Early termination/discontinuation.
Population: The analysis population included all participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07321332 (Suspension)/Ritonavir 300/100 mg BID, Fasted | Itraconazole 200 mg QD + PF-07321332(Suspension)/Ritonavir 300/100 mg BID, Fasted
Number analyzed (Participants) | 12 | 11
Participants
  PR interval, Aggregate (msec) Value >= 300 | 0 | 0
  PR interval, Aggregate (msec) %Change >= 25/50% | 0 | 0
  QRS Duration, Aggregate (msec) Value >= 140 | 0 | 0
  QRS Duration, Aggregate (msec) %Change >= 50% | 0 | 0
  QTcF interval, Aggregate (msec) 450 < Value < = 480 | 0 | 0
  QTcF interval, Aggregate (msec) 480 < Value < = 500 | 0 | 0
  QTcF interval, Aggregate (msec) Value > 500 | 0 | 0
  QTcF interval, Aggregate (msec) 30 < Change < = 60 | 0 | 0
  QTcF interval, Aggregate (msec) Change > 60 | 0 | 0

6. Secondary Outcome: Change From Baseline in Vital Signs Data - Supine Systolic Blood Pressure
Description: Vital signs(systolic and diastolic blood pressure, and pulse rate) were measured with participants after having a rest for at least 5 minutes in a supine position. Vital signs assessment were performed after collection of ECGs and prior to collection of blood draws if scheduled at the same time.
Time Frame: Screening up to Day 9 of Period 2 or Early termination/discontinuation.
Population: The analysis population included all participants who took at least 1 dose of study intervention.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | PF-07321332 (Suspension)/Ritonavir 300/100 mg BID, Fasted | Itraconazole 200 mg QD + PF-07321332(Suspension)/Ritonavir 300/100 mg BID, Fasted
Number analyzed (Participants) | 12 | 11
mmHg
  Period 1/Day 3 0 hour (H): number analyzed (Participants) | 11 | 0
  Period 1/Day 3 0 hour (H) | 1.4 (9.84) |
  Period 1/Day 3 1H 30min: number analyzed (Participants) | 11 | 0
  Period 1/Day 3 1H 30min | 1.5 (9.03) |
  Period 2/Day 4 0H: number analyzed (Participants) | 0 | 11
  Period 2/Day 4 0H |  | 2.6 (11.34)
  Period 2/Day6 0H: number analyzed (Participants) | 0 | 11
  Period 2/Day6 0H |  | 3.6 (8.43)
  Period 2/Day6 1H: number analyzed (Participants) | 0 | 11
  Period 2/Day6 1H |  | 5.5 (10.11)
  Period 2/Day6 1H 30min: number analyzed (Participants) | 0 | 11
  Period 2/Day6 1H 30min |  | 5.3 (13.52)
  Period 2/Day6 72 H: number analyzed (Participants) | 0 | 11
  Period 2/Day6 72 H |  | 6.4 (10.11)

7. Secondary Outcome: Change From Baseline in Vital Signs Data - Supine Diastolic Blood Pressure
Description: as for outcome 6
Time Frame: Screening up to Day 9 of Period 2 or Early termination/discontinuation.
Population: The analysis population included all participants who took at least 1 dose of study intervention.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | PF-07321332 (Suspension)/Ritonavir 300/100 mg BID, Fasted | Itraconazole 200 mg QD + PF-07321332(Suspension)/Ritonavir 300/100 mg BID, Fasted
Number analyzed (Participants) | 12 | 11
mmHg
  Period 1/Day 3 0H: number analyzed (Participants) | 11 | 0
  Period 1/Day 3 0H | -0.9 (4.97) |
  Period 1/Day 3 1H 30min: number analyzed (Participants) | 11 | 0
  Period 1/Day 3 1H 30min | 0.5 (4.74) |
  Period 2/Day 4 0H: number analyzed (Participants) | 0 | 11
  Period 2/Day 4 0H |  | 4.1 (4.09)
  Period 2/Day 6 0H: number analyzed (Participants) | 0 | 11
  Period 2/Day 6 0H |  | 3.5 (4.44)
  Period 2/Day 6 1H: number analyzed (Participants) | 0 | 11
  Period 2/Day 6 1H |  | 4.9 (4.87)
  Period 2/Day 6 1H 30min: number analyzed (Participants) | 0 | 11
  Period 2/Day 6 1H 30min |  | 4.2 (5.44)
  Period 2/Day 6 72H: number analyzed (Participants) | 0 | 11
  Period 2/Day 6 72H |  | 2.9 (6.28)

8. Secondary Outcome: Change From Baseline in Vital Signs Data - Supine Pulse Rate
Description: as for outcome 6
Time Frame: Screening up to Day 9 of Period 2 or Early termination/discontinuation.
Population: The analysis population included all participants who took at least 1 dose of study intervention.
Measure: Mean (Standard Deviation); unit: beats per minute(bpm)
Groups:
- PF-07321332 (Suspension)/Ritonavir 300/100 mg BID, Fasted 0/1: Participants received PF-07321332/ritonavir 300/100 mg administered orally every 12 hours for a total of 5 doses, from Day 1 morning to Day 3 morning of Period 1.
Arm/Group | PF-07321332 (Suspension)/Ritonavir 300/100 mg BID, Fasted 0/1 | Itraconazole 200 mg QD + PF-07321332(Suspension)/Ritonavir 300/100 mg BID, Fasted
Number analyzed (Participants) | 12 | 11
beats per minute(bpm)
  Period 1/Day 3 0 H: number analyzed (Participants) | 12 | 0
  Period 1/Day 3 0 H | -0.5 (5.92) |
  Period 1/Day 3 1 H 30 min: number analyzed (Participants) | 11 | 0
  Period 1/Day 3 1 H 30 min | -3.1 (4.64) |
  Period 2/Day 4 0 H: number analyzed (Participants) | 0 | 11
  Period 2/Day 4 0 H |  | -2.4 (5.50)
  Period 2/Day 6 0 H: number analyzed (Participants) | 0 | 11
  Period 2/Day 6 0 H |  | -2.5 (8.26)
  Period 2/Day 6 1 H: number analyzed (Participants) | 0 | 11
  Period 2/Day 6 1 H |  | -0.8 (10.84)
  Period 2/Day 6 1 H 30 min: number analyzed (Participants) | 0 | 11
  Period 2/Day 6 1 H 30 min |  | -2.1 (12.79)
  Period 2/Day 6 72 H: number analyzed (Participants) | 0 | 11
  Period 2/Day 6 72 H |  | 0.3 (9.96)

9. Secondary Outcome: Time for Cmax (Tmax) for PF-07321332
Description: PF-07321332 Tmax was observed directed from data
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hours(hr)
Arm/Group | PF-07321332 (Suspension)/Ritonavir 300/100 mg BID, Fasted | Itraconazole 200 mg QD + PF-07321332(Suspension)/Ritonavir 300/100 mg BID, Fasted
Number analyzed (Participants) | 11 | 11
hours(hr) | 1.020 [0.500 to 2.08] | 1.700 [0.500 to 4.00]

10. Secondary Outcome: Terminal Half-life(t1/2) of PF-07321332
Description: Terminal half-life was defined as the time measured for the plasma concentration of drug to decrease by one half.
Time Frame: as for outcome 1
Population: The analysis population included all participants who took at least 1 dose of study intervention and in whom at least 1 of the PK parameters of interest were reported. Here, "Number of Participants analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: hours(hr)
Arm/Group | PF-07321332 (Suspension)/Ritonavir 300/100 mg BID, Fasted | Itraconazole 200 mg QD + PF-07321332(Suspension)/Ritonavir 300/100 mg BID, Fasted
Number analyzed (Participants) | 11 | 10
hours(hr) | 8.255 (1.9465) | 7.793 (0.89019)

11. Secondary Outcome: Area Under the Plasma Concentration-time Profile From Time Zero to the Time of the Last Quantifiable Concentration(AUClast) of PF-07321332
Description: AUClast of PF-07321332 was determined by Linear/Log trapezoidal method.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-07321332 (Suspension)/Ritonavir 300/100 mg BID, Fasted | Itraconazole 200 mg QD + PF-07321332(Suspension)/Ritonavir 300/100 mg BID, Fasted
Number analyzed (Participants) | 11 | 11
ng*hr/mL | 41840 (21) | 74430 (21)

12. Secondary Outcome: Apparent Clearance(CL/F) of PF-07321332
Description: CL/F was apparent clearance.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | PF-07321332 (Suspension)/Ritonavir 300/100 mg BID, Fasted | Itraconazole 200 mg QD + PF-07321332(Suspension)/Ritonavir 300/100 mg BID, Fasted
Number analyzed (Participants) | 11 | 11
L/hr | 8.990 (20) | 6.478 (18)

13. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of PF-07321332
Description: Vz/F was apparent volume of distribution.
Time Frame: as for outcome 1
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | PF-07321332 (Suspension)/Ritonavir 300/100 mg BID, Fasted | Itraconazole 200 mg QD + PF-07321332(Suspension)/Ritonavir 300/100 mg BID, Fasted
Number analyzed (Participants) | 11 | 10
L | 104.7 (33) | 72.07 (16)

ADVERSE EVENTS:
Time Frame: From screening up to Day 35.
Description: Serious adverse events(SAE) and non-serious AEs were recorded on the case report form.
Arm/Group | PF-07321332 (Suspension)/Ritonavir 300/100 mg BID, Fasted | Itraconazole 200 mg QD + PF-07321332(Suspension)/Ritonavir 300/100 mg BID, Fasted
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 7/12 | 10/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-07321332 (Suspension)/Ritonavir 300/100 mg BID, Fasted (N=12) | Itraconazole 200 mg QD + PF-07321332(Suspension)/Ritonavir 300/100 mg BID, Fasted (N=11)
Atrioventricular block first degree (Cardiac disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 4
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Anorectal discomfort (Gastrointestinal disorders) | 0 | 1
Breath odour (Gastrointestinal disorders) | 1 | 3
Change of bowel habit (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 6
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Eructation (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Dysgeusia (Nervous system disorders) | 2 | 3
Headache (Nervous system disorders) | 4 | 3
Restless legs syndrome (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 1
Testicular pain (Reproductive system and breast disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Asthenia (General disorders) | 0 | 2
Fatigue (General disorders) | 1 | 2
Feeling hot (General disorders) | 0 | 1
Influenza like illness (General disorders) | 0 | 1
Injection site pain (General disorders) | 0 | 1
Vessel puncture site haematoma (General disorders) | 1 | 0
Vessel puncture site pain (General disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-07-02): https://cdn.clinicaltrials.gov/large-docs/22/NCT04962022/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-20): https://cdn.clinicaltrials.gov/large-docs/22/NCT04962022/SAP_001.pdf